CLINICAL TRIAL: NCT03488407
Title: A Prospective Study to Evaluate Feasibility of Routine Use of Radial Access for Primary Angioplasty and to Assess it in Subgroups With Unfavorable Characteristics
Brief Title: Evaluation of Feasibility of Radial Access for Primary Angioplasty and to Assess it in High Risk Subgroups
Status: Completed | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Dr Rajesh Sharma, Senior Resident, Jubilee Mission Medical College and Research Institute
Other Study IDs: 2/16/IEC/JMMC&RI
Record Dates: First submitted 2018-03-03; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Primary Angioplasty
Keywords: Primary angioplasty; Radial access; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary percutaneous coronary intervention is the preferred treatment for patients with ST-segment acute coronary syndrome. The radial access is an established approach, associated with a reduction in vascular access related complications after primary percutaneous coronary interventions. The purpose of this study is to examine the baseline characteristics, risk factors, procedural parameters and complications in patients with STEMI taken for primary angioplasty by radial access.

Data of all patients with acute STEMI with primary PCI through radial access is to be evaluated for baseline characteristics and procedural parameters and complications. Patients in the prospective study are followed up till discharge and any in-hospital complication noted.

This was a prospective, observational and descriptive study. Three hundred fifteen consecutive patients with an ST-segment elevation acute myocardial infarction (STEMI) treated with primary angioplasty by radial access, admitted between March 2016 and Feb 2017 were analyzed for their baseline characteristics, risk factors, and procedural parameters, complications and outcomes. High risk sub-groups analysis was also done. High risk groups includes patients with age >75yrs, cardiogenic shock, severe LV systolic dysfunction, acute left ventricular failure, high degree AV block, right ventricular infarction and low BMI. The study is conducted among patients with acute STEMI, considered for primary PCI through radial artery access at operator discretion.

This study analyzed the baseline characteristics of patients which includes clinical history, clinical examination, ECG, 2D ECHO, coronary angiogram to evaluate cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting with STEMI and being considered for primary PCI through radial access between March 2016 and Feb 2017.

Exclusion Criteria:

* Patients with ACS other than STEMI
* All primary PCI in STEMI through femoral access.
* All radial elective PCI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All prospective patients presenting with STEMI and being considered for primary PCI through radial access between March 2016 to Feb 2017.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2016-03-05 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of radial angioplasty success in whole cohort. | one year
  Angioplasty success rate (by TIMI flow grade)
Evaluation of in-hospital complication. | One year
  Rate of local complications

SECONDARY OUTCOMES:
High risk v/s non-high risk subgroup analysis | one year
  Non- inferiority of radial angioplasty for high risk group were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Sharma, MD, Principal Investigator — Jubilee Mission Medical College & Research Institute